CLINICAL TRIAL: NCT06128395
Title: Retrospective Study to Assess if Aspirin 162 mg is Better Than 81 mg for Embryo Transfer Outcomes
Brief Title: ASA 81 mg vs 162 mg During Frozen Embryo Transfer (FET)
Status: Completed | Type: Observational
Sponsor: Clinique Ovo (Industry)
Responsible Party: Sponsor
Other Study IDs: 3384
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Fertility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aspirin 81 mg for Frozen Embryo Transfer (FET): Subjects were prescribed Aspirin 81 mg to be started on the third day of their menstrual cycle in preparation for their FET.
  Interventions: Other: Frozen embryo transfer
- Aspirin 162 mg for Frozen Embryo Transfer (FET): Subjects were prescribed Aspirin 162 mg to be started on the third day of their menstrual cycle in preparation for their FET
  Interventions: Other: Frozen embryo transfer

INTERVENTIONS:
Other: Frozen embryo transfer — A frozen embryo transfer involves thawing a fertilized embryo and transferring it in the uterus in order to obtain a pregnancy

SUMMARY:
The use of low dose aspirin is recommended for high risk patients to reduce the risk of pre-eclampsia, placental abruption and antepartum hemorrhage. Recent studies have shown that in a specific population, the use of low dose aspirin might reduce the risk of preterm birth in pregnant women with singleton pregnancy. In June 2022, clinique ovo started implementing the use of Aspirin 162 mg instead of 81 mg in the frozen embryo transfer cycles based on recent study outcomes. The use of Aspirin 162 mg might have additional benefits on the embryo transfer outcomes by decreasing the miscarriage. Moreover this can be continued until late in pregnancy without adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* Women taking aspirin 81 mg or 162 mg prior to an autologous embryo transfer
* Age < 40 years old
* Embryo transfer cycle done at clinique ovo

Exclusion Criteria:

* Egg or embryo recipient
* History of recurrent miscarriages, defined as ≥ 3 consecutive losses
* Patients that needed Viagra, PRP or other modalities to improve their endometrial thickness
* Uterine factor infertility
* Abnormal hormonal profiles
* Stimulated embryo transfer cycles
* History of recurrent implantation failure defined as failed ≥ 2 euploid embryos transfer or ≥ 3 blastocysts

Max Age: 40 Years | Sex: Female
Age Groups: Child, Adult
Gender Based: Yes — Women able to have an embryo transfered in their uterus
Study Population: FET Data spreadsheet from January 2022 to December 2022
Sampling Method: Probability Sample
Enrollment: 1207 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-09-18 (Actual)

PRIMARY OUTCOMES:
Compare clinical pregnancy rate between patients prescribed Aspirin 81 mg vs Aspirin 162 mg | Time Frame: 6 to 8 weeks after Frozen Embryo Transfer
  clinical pregnancy is the presence of fetal heartbeat at the viability ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Wael Jamal, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No